CLINICAL TRIAL: NCT00887029
Title: A 12 Week Comparison of DuoTrav and Xalacom at 24 Hours Post-Dose in the Treatment of Open-Angle Glaucoma (the DVX Study)
Brief Title: A 12 Week Comparison of DuoTrav and Xalacom in Open-Angle Glaucoma
Acronym: DVX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ophthalmic Consultants Centres, Canada (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OCC1023
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Topical prostaglandin analogue; glaucoma; POAG; OHT; OAG; ocular hypertension; fixed combination protaglandin analogue therapy; DuoTrav; timolol; travoprost; 24 hour post dose; IOP; dosing preference
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Duotrav; Xalacom

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DuoTrav (Active Comparator)
  Interventions: Drug: DuoTrav (travoprost-timolol ophthalmic drops)
- Xalacom (Active Comparator)
  Interventions: Drug: Xalacom (latanoprost-timolol ophthalmic drops)

INTERVENTIONS:
Drug: DuoTrav (travoprost-timolol ophthalmic drops) — topical ophthalmic drops instilled 1 drop daily
  Other Names: DuoTrav
  Arms: DuoTrav
Drug: Xalacom (latanoprost-timolol ophthalmic drops) — topical ophthalmic drops instilled 1 drop daily
  Other Names: Xalacom
  Arms: Xalacom

SUMMARY:
Hypothesis:

* H1: Efficacy of Duotrav will be superior to Xalacom at 24 hours post dosing when both medications are given in the morning
* H2: A significant proportion of patients will prefer dosing of once daily topical fixed combination therapy in the morning compared to evening dosing

DETAILED DESCRIPTION:
* Primary objective: Compare IOP-lowering efficacy of morning dosing of Duotrav to Xalacom.
* Secondary objective: Compare patient dosing preferences for topical prostaglandin therapy in terms of convenience and perceived compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old, diagnosed with primary open angle glaucoma or ocular hypertension
* IOP currently uncontrolled on beta blocker monotherapy, as judged by the investigator
* Response to Timolol 0.5% was a ≥10% reduction in IOP
* IOP at 9:00 of ≥ 20 mmHg while still on beta blocker
* Non-prescription and prescription topical ophthalmic products and systemic medications other than those mentioned in the exclusion criteria will be allowed during the study.
* Patients wearing contact lenses will be permitted to participate in the study provided that the contact lenses are removed during instillation of study medication and that the patient waits fifteen (15) minutes following drug instillation to re-insert the lenses. Contact lenses cannot be worn on study days.

Exclusion Criteria:

* Best corrected visual acuity worse than 0.6 logMAR or 20/80 Snellen in either eye.
* Patients in whom the mean IOP in either eye at the screening exam visit is greater than 36 mmHg
* History of ocular trauma within the past six (6) months.
* History of ocular infection or ocular inflammation within the past three (3) months.
* History of chronic or recurrent severe inflammatory eye disease (i.e., scleritis, uveitis)
* History of severe or serious hypersensitivity to any components of the study medications.
* Any abnormality preventing reliable applanation tonometry of either eye.
* Intraocular surgery within the past six (6) months as determined by patient history and/or examination.
* Patients with cup/disc ratio greater than 0.80 in either eye.
* Patients with severe central visual field loss in either eye defined as a sensitivity 10 dB in at least two (2) of the four (4) visual field test points closest to the point of fixation.
* History of severe retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment.
* Current use of ANY glucocorticoid administered by any route. Patient must have washed out of the glucocorticoid for at least 4 weeks prior to study entry.
* Use of any systemic prostaglandin or prostaglandin analogue (e.g., CYTOTEC) within the last three months.
* Current use of topical non-steroidal anti inflammatory agents which inhibit cyclo-oxygenase and prostaglandin analogue synthesis.
* Any form of glaucoma other than open-angle glaucoma (with or without a pigment dispersion or pseudoexfoliation component).
* Current use of topical non-steroidal anti inflammatory agents which inhibit cyclo-oxygenase and prostaglandin analogue synthesis
* Angle grade less than 2 (extreme narrow angle with complete or partial closure) as measured by gonioscopy.
* Therapy with another investigational agent within the past 30 days
* Patients who would be at risk from treatment with a topical prostaglandin or prostaglandin analogue, are contraindicated for use of beta-blockers or any other medication used in this study, or who would be at risk from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
IOP lowering efficacy of DuoTrav and Xalacom | 12 weeks

SECONDARY OUTCOMES:
To compare patient dosing preferences in terms of convenience and perceived compliance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David B Yan, MD, Principal Investigator — Ophthalmic Consultant Centres; Navroop Gill, OD, Study Chair — Ophthalmic Consultant Centres
Locations (2):
- Canada (2):
  - Ophthalmic Consultant Centres, Mississauga, Ontario
  - Dr David B. Yan, M.D., F.R.C.S.C., Toronto, Ontario

REFERENCES:
- [Result] Netland PA, Landry T, Sullivan EK, Andrew R, Silver L, Weiner A, Mallick S, Dickerson J, Bergamini MV, Robertson SM, Davis AA; Travoprost Study Group. Travoprost compared with latanoprost and timolol in patients with open-angle glaucoma or ocular hypertension. Am J Ophthalmol. 2001 Oct;132(4):472-84. doi: 10.1016/s0002-9394(01)01177-1. PMID 11589866
- [Result] Dubiner HB, Sircy MD, Landry T, Bergamini MV, Silver LH, Darell Turner F, Robertson S, Andrew RM, Weiner A, Przydryga J. Comparison of the diurnal ocular hypotensive efficacy of travoprost and latanoprost over a 44-hour period in patients with elevated intraocular pressure. Clin Ther. 2004 Jan;26(1):84-91. doi: 10.1016/s0149-2918(04)90008-2. PMID 14996520
- [Result] Topouzis F, Melamed S, Danesh-Meyer H, Wells AP, Kozobolis V, Wieland H, Andrew R, Wells D. A 1-year study to compare the efficacy and safety of once-daily travoprost 0.004%/timolol 0.5% to once-daily latanoprost 0.005%/timolol 0.5% in patients with open-angle glaucoma or ocular hypertension. Eur J Ophthalmol. 2007 Mar-Apr;17(2):183-90. doi: 10.1177/112067210701700206. PMID 17415690
- [Result] Diestelhorst M, Larsson LI; European Latanoprost Fixed Combination Study Group. A 12 week study comparing the fixed combination of latanoprost and timolol with the concomitant use of the individual components in patients with open angle glaucoma and ocular hypertension. Br J Ophthalmol. 2004 Feb;88(2):199-203. doi: 10.1136/bjo.2003.018234. PMID 14736774
- [Result] Yan DB, Battista RA, Haidich AB, Konstas AG. Comparison of morning versus evening dosing and 24-h post-dose efficacy of travoprost compared with latanoprost in patients with open-angle glaucoma. Curr Med Res Opin. 2008 Nov;24(11):3023-7. doi: 10.1185/03007990802426813. Epub 2008 Oct 14. PMID 18826749
- [Result] Alm A, Stjernschantz J. Effects on intraocular pressure and side effects of 0.005% latanoprost applied once daily, evening or morning. A comparison with timolol. Scandinavian Latanoprost Study Group. Ophthalmology. 1995 Dec;102(12):1743-52. doi: 10.1016/s0161-6420(95)30798-1. PMID 9098273